CLINICAL TRIAL: NCT02042430
Title: A Pilot Study of the Immunological Effects of Neo-Adjuvant INCB024360 in Patients With Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Carcinoma
Brief Title: Epacadostat Before Surgery in Treating Patients With Newly Diagnosed Stage III-IV Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-02483; NCI-2013-02483 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ICD 10016180; CITN-05 OVARIAN IDO; ICD 10033159; ICD 10026669; CITN-05 (Other: Cancer Immunotherapy Trials Network); CITN-05 (Other: CTEP); P30CA015704 (NIH); U01CA154967 (NIH)
Record Dates: First submitted 2014-01-20; First posted 2014-01-22 (Estimated); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Stage III Fallopian Tube Cancer AJCC v7; Stage III Ovarian Cancer AJCC v6 and v7; Stage III Primary Peritoneal Cancer AJCC v7; Stage IIIA Fallopian Tube Cancer AJCC v7; Stage IIIA Ovarian Cancer AJCC v6 and v7; Stage IIIA Primary Peritoneal Cancer AJCC v7; Stage IIIB Fallopian Tube Cancer AJCC v7; Stage IIIB Ovarian Cancer AJCC v6 and v7; Stage IIIB Primary Peritoneal Cancer AJCC v7; Stage IIIC Fallopian Tube Cancer AJCC v7; Stage IIIC Ovarian Cancer AJCC v6 and v7; Stage IIIC Primary Peritoneal Cancer AJCC v7; Stage IV Fallopian Tube Cancer AJCC v6 and v7; Stage IV Ovarian Cancer AJCC v6 and v7; Stage IV Primary Peritoneal Cancer AJCC v7
MeSH Terms: conditions — Fallopian Tube Neoplasms | interventions — epacadostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (IDO1 inhibitor INCB024360) (Experimental): Patients receive IDO1 inhibitor INCB024360 PO BID on days 1-14 and undergo surgery on day 15. Treatment continues in the absence of disease progression or unacceptable toxicity. In circumstances where there are medical or administrative reasons for delaying surgery, treatment with IDO1 inhibitor INCB024360 may continue for up to 3 weeks.
  Interventions: Drug: Epacadostat; Other: Laboratory Biomarker Analysis; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Epacadostat — Given PO
  Other Names: INCB 024360; INCB024360
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Therapeutic Conventional Surgery — Undergo surgery

SUMMARY:
This pilot Early Phase I clinical trial studies epacadostat before surgery in treating patients with newly diagnosed stage III-IV epithelial ovarian, fallopian tube, or primary peritoneal cancer. Epacadostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the extent by which INCB024360 (epacadostat) alters the number of cluster of differentiation (CD)8+ T cells by immunohistochemistry (IHC).

SECONDARY OBJECTIVES:

I. To determine the extent by which INCB024360 alters the number and character of tumor infiltrating lymphocytes by IHC and gene signature by microarray analysis.

II. To determine the extent to which INCB024360 alters the character of the cellular content of peripheral blood mononuclear cells (PBMCs) and ascites fluid as determined by multiparameter flow cytometry.

III. To determine the extent to which INCB024360 alters PBMC and ascites fluid transcriptomes.

IV. To determine whether INCB024360 alters the ongoing and nascent anti-tumor responses antigens associated with ovarian cancer (e.g., cancer/testis antigen 1B [NY-ESO-1], preferentially expressed antigen in melanoma [PRAME] and mesothelin) as well as memory viral responses (influenza A), and chronic viral responses (cytomegalovirus).

V. To assess the safety and tolerability of INCB024360. VI. To determine the extent to which a regimen of INCB024360 that normalizes serum kynurenine/tryptophan (Kyn/Trp) ratios will alter the tumor microenvironment by assessing the ascites and intra-tumor Kyn/Trp ratios at the time of surgery, one day after stopping INCB024360.

VII. To associate any observed changes with the expression of IDO1 protein by IHC in tumor or tumor infiltrating cells.

OUTLINE:

Patients receive epacadostat orally (PO) twice daily (BID) on days 1-14 and undergo surgery on day 15. Treatment continues in the absence of disease progression or unacceptable toxicity. In circumstances where there are medical or administrative reasons for delaying surgery, treatment with epacadostat may continue for up to 3 weeks.

After completion of study treatment, patients are followed up for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed stage III or IV epithelial ovarian, fallopian or primary peritoneal carcinoma with or without ascites and potentially resectable disease agreeing to debulking surgery as standard therapy
* Pre-surgery tumor deemed amenable to core biopsy (with at least 100 mm^3 tumor volume per biopsy)
* Patients must be willing and able to undergo ascites fluid collection pre- and post-study treatment if adequate ascites is present; patients without adequate ascites may also participate in the trial
* Patients must be willing and able to undergo a pre-surgery biopsy and wait 2 weeks before their debulking surgery; NOTE: consented patients with subsequent inadequate biopsy material will not receive INCB024360 or be analyzed and will be replaced; the study will be stopped if adequate tissue is not obtained in more than 2/3 of paired samples with a maximum accrual of 18 patients
* Women of all races and ethnic groups are eligible for this trial
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 (Karnofsky > 70%)
* Any human leukocyte antigen (HLA) type
* Life expectancy of at least 6 months
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,000/mcL
* Platelets >= 100,000/mcL
* Hemoglobin > 11g/dL
* Total bilirubin < 1.5 x institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) up to 2.5 times upper limit of normal (ULN)
* Creatinine < 1.5 x institutional upper limit of normal OR creatinine clearance > 60 ml/min OR > 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Prothrombin time (PT), international normalized ratio (INR) less than 1.5 times the institutional upper limit of normal
* Females of childbearing potential must have a negative pregnancy test within 48 hours prior to initiation of protocol therapy; women of child-bearing potential must agree to use adequate contraception prior to study entry and for the duration of study participation, and 4 months after completion of INCB024360; effective birth control includes (a) intrauterine device (IUD) plus one barrier method; or (b) 2 barrier methods; effective barrier methods are male or female condoms, diaphragms, and spermicides (creams or gels that contain a chemical to kill sperm) (c) oral contraceptive pills and (d) intramuscular DEPO medroxyprogesterone acetate; should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately

  * NOTE: subjects are considered not of childbearing potential if they are surgically sterile, they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy or they are postmenopausal; menopause is the age associated with complete cessation of menstrual cycles, menses, and implies the loss of reproductive potential; by a practical definition, it assumes menopause after 1 year without menses with an appropriate clinical profile at the appropriate age
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had prior systemic therapy or radiotherapy for stage III or IV epithelial ovarian, fallopian or primary peritoneal carcinoma
* Extensive active brain disease including symptomatic brain metastases or presence of leptomeningeal disease
* Concomitant systemic treatment with corticosteroids, anti-histamine or non-steroidal anti-inflammatory drugs; any cyclooxygenase-2 (COX-2) inhibitors are permitted
* Use of any UDP glucuronosyltransferase 1 family, polypeptide A9 (UGT1A9) inhibitor including: acitretin, amitriptyline, androsterone, cyclosporine, dasatinib, diclofenac, diflunisal, efavirenz, erlotinib, estradiol (17-beta), flutamide, gefitinib, gemfibrozil, glycyrrhetinic acid, glycyrrhizin, imatinib, imipramine, ketoconazole, linoleic acid, mefenamic acid, mycophenolic acid, niflumic acid, nilotinib, phenobarbital, phenylbutazone, phenytoin, and probenecid propofol, quinidine, ritonavir, sorafenib, sulfinpyrazone, valproic acid, and verapamil; patients must avoid UGT1A9 inhibitors from the screening period through active treatment with INCB024360 and for one week after discontinuation of INCB024360
* Uncontrolled intercurrent illness including, but not limited to:

  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Congestive heart failure
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Medical or psychiatric illness that would, in the opinion of the investigator, preclude participation in the study or the ability of patients to provide informed consent for themselves
* Pregnancy or nursing or unwilling to take adequate birth control during therapy; NOTE: breastfeeding should be discontinued
* Known human immunodeficiency virus (HIV) or other history of immunodeficiency disorder
* Patients who had, within the past 6 months, a cardiovascular accident (CVA) or at risk for arterial thrombus such as severe peripheral vascular disease (PVD) and carotid artery disease (CAD)
* History of autoimmune disorders requiring cytotoxic or immunosuppressive therapy, or autoimmune disorders with visceral involvement; active or inactive auto-immune disorders (e.g., rheumatoid arthritis, moderate or severe psoriasis, multiple sclerosis, systemic lupus erythematosus, inflammatory bowel disease, etc.) requiring treatment

  * The following will not be exclusionary:

    * Vitiligo, thyroiditis or eczema requiring systemic steroids at a dose =< 7.5 mg/day of prednisone or equivalent; individual cases can be discussed with the principal investigator
* History of pulmonary disease such as emphysema or chronic obstructive pulmonary disease (COPD), (forced expiratory volume of the lung in 1 second [FEV1] > 60% of predicted for height and age); pulmonary function tests (PFTs) are required in patients with prolonged smoking history or signs, symptoms, or history of respiratory dysfunction)
* Cirrhosis or chronic hepatitis C virus positivity or chronic hepatitis B infection; subjects who may not tolerate immune-mediated hepatitis due to compromised hepatic reserve are also excluded from participation including: 1) subjects with extensive liver metastasis (as judged by the investigator) 2) subjects who drink more than two standard alcoholic beverages per day on a regular basis 3) subjects who consume more than 2 grams of acetaminophen per day on a regular basis

  * A positive hepatitis B serology indicative of previous immunization (i.e., hepatitis B surface antibody [HBsAb] positive and hepatitis B core antibody [HBcAb] negative), or a fully resolved acute hepatitis B virus (HBV) infection is not an exclusion criterion
* Concurrent systemic immunosuppressive therapy or steroid therapy with more than 7 consecutive days of steroids within the last 4 weeks

  * The use of prednisone or equivalent < 0.125 mg/kg/day (absolute maximum of 10 mg/day) as replacement therapy is permitted
  * Inhaled corticosteroids are permitted
  * The following will not be exclusionary:

    * The presence of laboratory evidence of autoimmune disease (e.g. positive antinuclear antibody [ANA] titer) without associated symptoms
    * Mild Raynaud's phenomenon
    * History of severe asthma, as defined by prior or current use of systemic corticosteroids for disease control, with the exception of physiological replacement doses of cortisone acetate or equivalent, as defined by a dose of prednisone or equivalent of 10 mg or less
* Malabsorption syndrome or chronic nausea that might hinder absorption and assessment of oral medication
* Cardiovascular disease that meets one of the following: congestive heart failure (New York Heart Association class III or IV), active angina pectoris, or recent myocardial infarction (within the last 6 months)
* History of pulmonary embolus and/or substantial deep vein thrombosis
* Patient with prior malignancies other than ovarian cancer for which the patient has not been disease free for 3 years or more, except treated and cured basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix
* Therapy with monoamine oxidase inhibitors (MAOIs) and selective serotonin reuptake inhibitor (SSRIs) within the last 4 weeks or history of serotonin syndrome
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or medical (e.g. infectious) illness
* Any underlying medical or psychiatric condition, which in the opinion of the investigator, will make the administration of INCB024360 hazardous or obscure the interpretation of adverse events
* Unable or unwilling to swallow tablets BID
* Subjects with any concurrent condition that, in the investigator's opinion, would jeopardize the safety of the subject or compliance with the protocol
* Low-dose Coumadin (1 mg) is acceptable; however, doses that increase INR are not permitted; if an alternative to Coumadin-based anticoagulants cannot be used, the INR should be monitored weekly after initiation of therapy and upon discontinuation of INCB024360, until INR normalization

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-08-25 (Actual); Primary Completion 2016-11-29 (Actual); Study Completion 2016-11-29 (Actual)

PRIMARY OUTCOMES:
Number of participants with an increase in CD8+ T cells | Baseline to day 15
  The correlation between results of the IDO expression levels analyzed by IHC and the Kyn/Trp ratios will be analyzed if available.

SECONDARY OUTCOMES:
Change in number and character of tumor infiltrating lymphocytes | Baseline to up to day 35
Change in gene signatures as assessed by microarray analysis | Baseline to up to day 35
Change in character of the cellular content of PBMCs and ascites fluid, determined by multiparameter flow cytometry | Baseline to up to day 35
Change in fluid transcriptomes in PBMC and ascites | Baseline to up to day 35
Change in ongoing and nascent anti-tumor response antigens associated with ovarian cancer, including NY-ESO-1, PRAME and mesothelin | Baseline to up to day 35
Change in memory viral responses, including influenza A | Baseline to up to day 35
Change in chronic viral responses, including cytomegalovirus | Baseline to up to day 35
Incidence of adverse events, assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 1 year
Kyn/Trp ratios | Day 15
Changes in IDO1 expression by IHC | Baseline to up to day 35

CONTACTS AND LOCATIONS:
Overall Officials: Kunle Odunsi, Principal Investigator — Cancer Immunotherapy Trials Network
Locations (2):
- United States (2):
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Roswell Park Cancer Institute, Buffalo, New York